CLINICAL TRIAL: NCT06459635
Title: Prediction Study of the Pain Phase of Migraine Attacks in Patients With Episodic Migraine
Brief Title: Migraine Attack Pain Phase Prediction Study
Acronym: PREDI-CRISIS
Status: Recruiting | Type: Observational
Sponsor: Fundación de Investigación Biomédica - Hospital Universitario de La Princesa (Other)
Collaborators: Hospital Vall d'Hebron (Other); Hospital Donostia (Other); Hospital Universitario Marqués de Valdecilla (Other); Hospital Clínico Universitario Lozano Blesa (Other); Hospital Universitario La Fe (Other); Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Sponsor
Other Study IDs: 3513
Record Dates: First submitted 2024-06-05; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-06

CONDITIONS: Migraine; Migraine Headache; Migraine Disorders; Migraine Without Aura; Migraine With Aura
Keywords: Migraine; Headache; Predict; Prediction; headache prediction; predict headache; migraine prediction; predict migraine; migraine attacks; migraine attack; headache attack; migraine attack prediction; predict migraine attack; prediction algorithm; algorithm
MeSH Terms: conditions — Migraine Disorders; Migraine without Aura; Migraine with Aura; Headache

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with episodic migraine: Patients with episodic migraine who present between 4 and 10 migraine attacks per month. These patients must have a diagnosis of migraine by a headache neurologist and according to the criteria proposed by ICHD-3. In addition, they must present at least 1 year of evolution of the migraine, as well as a normal neurological examination and have given their informed consent.
- Control patients: People who have never had a headache episode with migraine characteristics. These may present, at most, one episode per month of headache with non-migraine characteristics in the last 3 months. In turn, they should not have a family history of migraine (1st and 2nd degree).

SUMMARY:
The study of the ability to predict pain in a migraine attack, through premonitory symptoms and through an ambulatory monitoring device through real-time recording of hemodynamic variables, is one of the strategic lines of research of the unit. of Headaches at the Hospital de La Princesa since 2013 together with the Complutense and Polytechnic University of Madrid. Their results have been reflected in various publications (Pagán J, et al. Sensors 2015; Gago-Veiga AB, et al. J Pain Res 2018) and have promoted the creation of several invention patents.

DETAILED DESCRIPTION:
Patients with episodic migraine will be recruited from the monographic headache clinics of the 7 centers participating in the study. These patients, for a maximum period of 2 months, must monitor their hemodynamic variables with a wearable device and record all the clinical characteristics of their migraine attacks. Subsequently, with these records, an individualized algorithm will be created for each patient that aims to predict the onset of the migraine attack.

ELIGIBILITY:
Inclusion Criteria:

* Age between 15 years and 69 years.
* Diagnosed with migraine by a headache neurologist and according to the criteria proposed by ICHD-3.
* History of migraine of at least 1 year of evolution.
* Normal neurological examination.
* Have given your informed consent.
* Be able to describe your clinical situation and the characteristics of your headache.
* Have an average of 10 to 14 migraine days per month in the three months prior to inclusion (high-frequency episodic migraine).
* User-level management capacity of "smartphone" type electronic devices.
* Be able to complete two months of study follow-up.

Exclusion Criteria:

* Presence of another type of headache, with the exception of headache due to excessive use of analgesic medication.
* Cognitive deficiency or any other pathology that may prevent or make it difficult for the patient to perform the study correctly.
* Neurological focus in the examination.
* Pregnancy or breastfeeding period.
* Patients with known heart disease or bronchopathy, Sjögren's syndrome, diabetes mellitus, or hypo/hyperthyroidism.
* Carriers of pacemakers, neurostimulators or any other electronic device that is considered to make the interpretation of biometric records difficult.
* Anatomical problem that makes the use of the device impossible.
* Patients in whom it is expected that a change in migraine preventive treatment or other usual treatment will be possible during the study period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients aged between 18 and 65 years with a diagnosis of episodic migraine who have between 4 and 14 days of headache per month. These patients will come from 7 Headache Units in Spain belonging to the following hospitals: • La Princesa University Hospital • Vall 'Hebron University Hospital • Marqués de Valdecilla University Hospital • Valladolid University Clinical Hospital • Donostia University Hospital • Lozano Blesa University Clinical Hospital • La Fe Polytechnic University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Development of a prediction strategy for the onset of migraine | From the beginning of treatment, which is the initial visit, to 2 months of follow-up
  Develop a prediction strategy for the onset of migraine attacks in patients with episodic migraine, based on hemodynamic and clinical variables of migraine attacks.

SECONDARY OUTCOMES:
Posibility of predict the onset of pain in a migraine attack | From the beginning of treatment, which is the initial visit, to 2 months of follow-up
  To analyze whether it is possible to predict the onset of pain in a migraine attack, through ambulatory and non-invasive monitoring of physiological variables.
Individualized prediction algorithm | From the beginning of treatment, which is the initial visit, to 2 months of follow-up
  Implement an individualized prediction algorithm that allows real-time prediction of the symptomatic phase of the migraine attack.
Effectiveness of the prediction model | From the beginning of treatment, which is the initial visit, to 2 months of follow-up
  Measure the effectiveness of the prediction model both at the individual level and in a large group of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Beatriz Gago Veiga, Principal Investigator — Fundación de Investigación Biomédica - Hospital Universitario de La Princesa
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Anonymized data may be shared upon reasonable request to the principal investigator.

REFERENCES:
- [Result] Gago-Veiga AB, Pagan J, Henares K, Heredia P, Gonzalez-Garcia N, De Orbe MI, Ayala JL, Sobrado M, Vivancos J. To what extent are patients with migraine able to predict attacks? J Pain Res. 2018 Sep 27;11:2083-2094. doi: 10.2147/JPR.S175602. eCollection 2018. PMID 30310310
- [Result] Pagan J, De Orbe MI, Gago A, Sobrado M, Risco-Martin JL, Mora JV, Moya JM, Ayala JL. Robust and Accurate Modeling Approaches for Migraine Per-Patient Prediction from Ambulatory Data. Sensors (Basel). 2015 Jun 30;15(7):15419-42. doi: 10.3390/s150715419. PMID 26134103